CLINICAL TRIAL: NCT02845960
Title: The Influence of Rapid Recovery on Sleep Quality Following Total Knee Replacement Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Yang, Professor, Southwest Hospital, China
Other Study IDs: Southwest Hospital
Record Dates: First submitted 2016-07-23; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Arthroplasty, Replacement, Knee; Recovery of Function; Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental group: rapid recovery
  Interventions: Behavioral: rapid recovery
- Controlled group: no rapid recovery

INTERVENTIONS:
Behavioral: rapid recovery — rapid recovery
  Groups: Experimental group

SUMMARY:
The purpose of this study is to evaluate the influence of rapid recovery on sleep quality following total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Primary unilateral total knee artropasty;
2. Patients with Knee osteoartritis or Rheumatoid arthritis;
3. Able and willing to provide signed informed consent.

Exclusion Criteria:

1. Simultaneously bilateral total knee artropasty or revision case;
2. Surgical History of the knee joint;
3. Knee joint cavity paracentesis in recent 3 months;
4. Stiffness with knee;
5. Blood coagulation disorders;
6. History of deep venous thrombosis;
7. Concomitant medical problems such as uncontrolled hypertention, severe cardiovascular disorder, chronic obstructive pulmonary disease, liver or renal failure
8. allergic to NSAIDs, opioid analgesics, zolpidem
9. sleep apnea, Parkinson disease, dementia, depression
10. use of sedatives or hypnotics
11. inability to comply with polysomnographic measurement

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
WOMAC score | 1 mounth
GAD-7 | 1 mounth
PSQI index | 1 mounth
Insomnia severity index | 1 mounth
polysomnographic measurement | 1 mounth
VAS | 1 mounth
Range of motion | 1 mounth

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No